CLINICAL TRIAL: NCT06056466
Title: A Prospective, Observational, Non-interventional, Single-center Study to Analyze the Relationship Between Different Vascular and Renal Parameters in Living Kidney Donors With 1 Year Follow-up
Brief Title: Different Vascular and Renal Parameters in Living Kidney Donors
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: CRC2018Tx
Record Dates: First submitted 2023-07-14; First posted 2023-09-28 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Renal Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic kidney disease (CKD) has a high prevalence globally and is a global health concern. CKD is associated with increased risks of cardiovascular morbidity, mortality and therefore decreased quality of life in any stage of the disease. CKD in early stage is often asymptomatic, which makes the detection of the disease difficult.

In this study our goal is to analyze in a clinical trial to what extend renal and vascular parameters correlate with histological kidney changes, especially in a population with eGFR rate of more than 60 mL/min/1.73 m² or pseduonormalized renal function. Our crossectional analysis focus on the association of abnormal vascular and renal parameters with histological renal changes. Our longitudinal analysis focus on the association of histological with renal and/or vascular parameters at baseline, with the renal outcome after kidney donation.

Different renal and vascular parameters are obtained non-invasively in potential living kidney donors before donation. Preimplantation kidney biopsies are obtained routinely during donation, which is a standard procedure of our living kidney donation programme. The living kidney donors will be followed up in respect to renal function and blood pressure for one year after donation.

Our hypothesis is that histological scoring of renal damage (total renal chronicity scores) correlates with vascular parameters indicating increased stiffness. The primary vascular parameter is wall to lumen ratio of retinal arterioles. Moreover the investigators hypothesize that vascular parameters predicts 24-hour blood pressure and renal outcome (eGFR, albuminuria) one year after donation. To prove this hypothesis overall the investigators will include 25 subjects in this study, having been evaluated before as potential living kidney donors. Total duration of this study for each volunteer is 15 months with total 5 visits, of which 4 are at the Clinical Research Unit (CRC) of the Department of Nephrology, University of Erlangen-Nuremberg and one is the day of kidney donation.

This study is important to detect renal damage or CKD in patients with eGFR rate of more than 60 mL/min/1.73 m² or pseduonormalized renal function (CKD stage 1 or 2).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) has a high prevalence globally and is a global health concern. KDIGO-Guidelines describes CKD as an abnormality of kidney function or structure, present more than 3 months, with implications for the health of an individual. CKD is associated with increased risks of cardiovascular morbidity, mortality and decreased quality of life in all stages of the disease. Most patients with CKD will die of cardiovascular event in earlier stages before end-stage renal disease develops. CKD in early stage is often asymptomatic, which makes the detection of the disease difficult. Early detection of CKD could delay or even prevent the associated complications and the progression to kidney failure through appropriate control of cardiovascular risk factors.

The glomerular filtration rate (GFR) is widely accepted as an overall index of kidney function and is considered for the classification of CKD. A GFR rate of more than 60 mL/min/1.73 m² is considered only as abnormal, if it is accompanied by albuminuria, urine sediment abnormalities, structural abnormalities detected by imaging tests, or if the patient has had a kidney biopsy with histological abnormalities. Since kidney biopsy is not done in all patients with respect to risk of the procedure, diagnosis of CKD stage 1 and 2 is difficult.

Moreover, an association of abnormal increase in GFR with all-cause mortality has also been recently described. This process of glomerular hyperfiltration may lead to pseudonormalization of the renal function and is associated with various medical conditions such as diabetes, hypertension as well as lifestyle factors, such as smoking and lack of physical activity. The influence of intrauterine environment in the development of low nephron number, leading to glomerular hyperfiltration and glomerular enlargement has been also described. These maladaptive changes may then eventually lead to the development of glomerular and systemic hypertension and renal disease in later life.

In this study our goal is to analyze in a clinical trial to what extend renal and vascular parameters correlate with histological kidney changes, especially in subjects with eGFR rate of more than 60 mL/min/1.73 m² or pseduonormalized renal function. Different renal and vascular parameters are obtained non-invasively in potential living kidney donors before donation. Kidney biopsies are obtained routinely after nephrectomy and before implantation (pre-implantation biopsy). Kidney biopsy samples can demonstrate definitive evidence of CKD through common histological changes. Our crosssectional analysis focus on the association of abnormal vascular and renal parameters with histological renal changes. The living kidney donors will be followed up in respect to renal function and blood pressure for one year after donation. Our longitudinal analysis focus on the association of histological with renal and/or vascular parameters at baseline, with the renal outcome (eGFR, albuminuria, 24-hour blood pressure) after kidney donation.

This study is a single-centre clinical study with 25 potential kidney donors. This is an exploratory and non-confirmatory study, in which the investigators analyse different vascular and renal parameters in potential kidney donors before donation and a kidney biopsy sample is obtained during donation.

Our hypothesis is that histological scoring of renal damage (total renal chronicity scores) correlates with vascular parameters indicating increased stiffness. The primary vascular parameter is wall to lumen ratio of retinal arterioles. Moreover the investigators hypothesize that vascular parameters predicts 24-hour blood pressure and renal outcome (eGFR, albuminuria) one year after donation.

This study is a single-center clinical study at the Clinical Research Unit (CRC) of the Department of Nephrology and Hypertension (Erlangen, Ulmenweg 18, 91054 Erlangen (INZ, University Hospital Erlangen)).

After approval of the trial protocol by the local ethics committee (University of Erlangen-Nuremberg), participants will be recruited from the transplantation center of Erlangen-Nuremberg, Germany. Eligible participants will be screened according to the inclusion and exclusion criteria on Visit 1 after approval of donation by immunological, psychological, medical evaluation and positive vote of the living donation commission. Subsequently suitable participants will be included in the trial after written informed consent has been obtained. The trial will be conducted in accordance with the Declaration of Helsinki and the principles of good clinical practice guidelines.

Demographic data, safety parameters (e.g. creatinine, liver enzymes), ECG and urine examination are obtained on visit 1. On the same day office BP and heart rate measurements are taken in a seated position after 5 min of rest according to guideline recommendations.

On visit 2 the subjects will be instructed to fast and abstain from alcohol, caffeine and antioxidant vitamins. The primary objective of this trial will be obtained on visit 2 in 25 potential kidney donors. On visit 2 vascular assessment including pulse wave analysis and velocity as well as flow mediated dilation (FMD) measurement will be performed. Retinal capillary flow (RCF) and structural and functional vascular changes of retinal arterioles will be assessed by Scanning Laser Doppler Flowmetry (SLDF) measurement. Resistance index of intrarenal arteries will be determined by renal duplex sonography. In patients without contraindications for MRI examination, ASL-MRI and 23Na-MRI will be performed on the same day. Blood samples will be drawn after lying half an hour in supine position to analyse renal (eGFR, Cystatin C) and endocrine (renin, angiotensin, aldosterone) parameters. Urine samples will be collected to assess UACR. At the end of visit a container will be handed over to the subject to collect urine for 24 hours to assess UACR, sodium, potassium and creatinine.

On the day of kidney donation (visit 3) a kidney biopsy sample will be obtained after explantation of the kidney, which is a standard procedure of our living kidney donor programme. Histological analysis and scoring of chronic changes such as global and segmental glomerulosclerosis, tubular atrophy, interstitial fibrosis and arteriosclerosis/arteriolosclerosis of the biopsy specimen will be performed.

The living kidney donors will be followed up according to our standard living kidney post-donation programme (visit 4 and 5) in respect to renal function (eGFR [CKD-Epi], Cystatin C, UACR), blood pressure (office and 24h ambulatory blood pressure) and endocrine parameters (renin, angiotensin, aldosterone) for one year after donation. If feasible, 24h-urine will be collected to re-assess parameters mentioned above. All assessments measured at visit 2 except measurement of FMD and measurement of resistance index of intrarenal arteries will be remeasured at visit 4. Safety parameters and adverse events will be recorded at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Age of 30 - 85 years
* Male and Female patients
* Persons (evaluated and accepted for kidney donation) in good and stable health condition with eGFR>60 ml/min/1.73m²
* Informed consent has to be given in written form

Exclusion Criteria:

* Type-2-diabetes or any other form of diabetes (fasting plasma glucose ≥ 126 mg/dl, HbA1c ≥ 6,5%, post prandial glucose ≥ 200 mg/dl *
* Uncontrolled arterial hypertension (≥ 180/110 mmHg) *
* Any history of stroke, transient ischemic attack, instable angina pectoris or myocardial infarction within the last 6 months prior to study inclusion *
* Estimated glomerular filtration rate ≤ 60 ml/min/1.73m² *
* Significant laboratory abnormalities such as Serum Glutamate-Oxaloacetate-Transaminase (SGOT) or Serum Glutamate-Pyruvate-Transaminase (SGPT) levels more than 3 times above the upper limit of normal range *
* Patients in unstable conditions due to any kind of serious disease, that infers with the conduction of the trial *
* Patients suffering from cataract or glaucoma +
* Diabetic retinopathy *
* active Drug or alcohol abuse *
* Pregnant and breast-feeding patients *
* Body mass index > 33 kg/m² *
* Participation in another clinical study within 30 days prior to visit 1+
* Subjects who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V +

For patients undergoing 23Na- and ASL-MRI:

* Implanted pacemakers or defibrillators +
* Other implanted metallic devices, which are not MRI compatible +
* Claustrophobia +
* Any other relevant clinical contraindication of MRI examination +

  * Please note that these exclusion criteria are also exclusion criteria of our kidney donation programme + These exclusions are due to the study, in particular due to methods we apply at visit 2

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the transplantion center of Erlangen-Nuremberg, Germany. Eligible participants will be screened according to the inclusion and exclusion criteria on Visit 1 after approval of donation by immunological, psychological, medical evaluation and positive vote of the living donation commission.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Wall to lumen ratio of retinal arterioles assessed by SLDF | within 8 weeks before donation, 6 months after donation
  The primary objective of the study is to analyze wall to lumen ratio of retinal arterioles before kidney donation and 6 months after donation

SECONDARY OUTCOMES:
Retinal capillary flow determined by SLDF measurement | within 8 weeks before donation, 6 months after donation
  change in retinal capillary flow 6 months after kidney donation
Central systolic pressure assessed by Sphygmocor XCEL | within 8 weeks before donation, 6 months after donation
  change in central systolic pressure 6 months after kidney donation
Pulse pressure assessed by Sphygmocor XCEL | within 8 weeks before donation, 6 months after donation
  change in pulse pressure 6 months after kidney donation
Pulse wave velocity assessed by Sphygmocor XCEL | within 8 weeks before donation, 6 months after donation
  change in pulse wave velocity 6 months after kidney donation
Augmentation index assessed by Sphygmocor XCEL | within 8 weeks before donation, 6 months after donation
  change in augmentation index 6 months after kidney donation
24-h ambulatory vascular parameter assessed by Mobil-O-Graph | within 8 weeks before donation, 6 months after donation, 1 year after donation
  change of 24-h ambulatory vascular parameter (pulse wave velocity) 6 months and 1 year after kidney donation
Flow mediated vasodilation as measured by semi-automated ultrasound system (% vasodilation from baseline) with the UNEX system | within 8 weeks before donation, 6 months after donation
  change of flow mediated vasodilation 6 months after kidney donation
Renal perfusion of both kidneys assessed by Arterial Spin Labeling MRI | within 8 weeks before donation, 6 months after donation
  change of renal perfusion (total, cortical, medullary) 6 months after kidney donation
Skin sodium content (23Na-MRI) assessed at the lower leg | within 8 weeks before donation, 6 months after donation
  change of Skin sodium content 6 months after kidney donation
Muscle sodium content (23Na-MRI) assessed at the lower leg | within 8 weeks before donation, 6 months after donation
  change of muscle sodium content 6 months after kidney donation
Resistance index determined by renal duplex sonography | within 8 weeks before donation, 6 months after donation
  change of resistance index 6 months after kidney donation
24-h ambulatory blood pressure assessed by Mobil-O-Graph | within 8 weeks before donation, 6 months after donation, 1 year after donation
  change of 24-h blood pressure 6 months and 1 year after kidney donation
estimated glomerular filtration rate (CKD-Epi) assessed in our central lab | within 8 weeks before donation, 6 months after donation, 1 year after donation
  change of estimated glomerular filtration rate (CKD-Epi) 6 months and 1 year after kidney donation
Cystatin C assessed in our central lab | within 8 weeks before donation, 6 months after donation, 1 year after donation
  change of Cystatin C 6 months and 1 year after kidney donation
UACR in spot urine and 24-h urine assessed in our central lab | within 8 weeks before donation, 6 months after donation, 1 year after donation
  change of UACR 6 months and 1 year after kidney donation
Global and segmental glomerulosclerosis (histological analyses of the kidney sample) | within 8 weeks after assessing primary outcome measure
  Global and segmental glomerulosclerosis analyzed histologically in a kidney biopsy sample obtained after explantation of the kidney.
  Minimum value=0, maximum value=3. Subjective histological assessment based on grade of glomerular sclerosis.
Tubular atrophy (histological analyses of the kidney sample) | within 8 weeks after assessing primary outcome measure
  Tubular atrophy analyzed histologically in a kidney biopsy sample obtained after explantation of the kidney.
  Minimum value=0, maximum value=3. Subjective histological assessment based on grade of tubular atrophy.
Interstitial fibrosis (histological analyses of the kidney sample) | within 8 weeks after assessing primary outcome measure
  Interstitial fibrosis analyzed histologically in a kidney biopsy sample obtained after explantation of the kidney.
  Minimum value=0, maximum value=3. Subjective histological assessment based on grade of fibrosis.
Arteriosclerosis/arteriolosclerosis (histological analyses of the kidney sample) | within 8 weeks after assessing primary outcome measure
  Arteriosclerosis/arteriolosclerosis analyzed histologically in a kidney biopsy sample obtained after explantation of the kidney.
  Minimum value=0 (Intima thickness less than thickness of media), maximum value=1 (Intima thickness greater than thickness of media)
Total renal chronicity score (histological analyses of the kidney sample) | within 8 weeks after assessing primary outcome measure
  Total renal chronicity score assessed histologically after explantation of the kidney.
  Minimum value=0 (better outcome), maximum value=10 (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill NR, Fatoba ST, Oke JL, Hirst JA, O'Callaghan CA, Lasserson DS, Hobbs FD. Global Prevalence of Chronic Kidney Disease - A Systematic Review and Meta-Analysis. PLoS One. 2016 Jul 6;11(7):e0158765. doi: 10.1371/journal.pone.0158765. eCollection 2016. PMID 27383068
- [Background] Eckardt KU, Coresh J, Devuyst O, Johnson RJ, Kottgen A, Levey AS, Levin A. Evolving importance of kidney disease: from subspecialty to global health burden. Lancet. 2013 Jul 13;382(9887):158-69. doi: 10.1016/S0140-6736(13)60439-0. Epub 2013 May 31. PMID 23727165
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Perlman RL, Finkelstein FO, Liu L, Roys E, Kiser M, Eisele G, Burrows-Hudson S, Messana JM, Levin N, Rajagopalan S, Port FK, Wolfe RA, Saran R. Quality of life in chronic kidney disease (CKD): a cross-sectional analysis in the Renal Research Institute-CKD study. Am J Kidney Dis. 2005 Apr;45(4):658-66. doi: 10.1053/j.ajkd.2004.12.021. PMID 15806468
- [Background] Keith DS, Nichols GA, Gullion CM, Brown JB, Smith DH. Longitudinal follow-up and outcomes among a population with chronic kidney disease in a large managed care organization. Arch Intern Med. 2004 Mar 22;164(6):659-63. doi: 10.1001/archinte.164.6.659. PMID 15037495
- [Background] Park M, Yoon E, Lim YH, Kim H, Choi J, Yoon HJ. Renal hyperfiltration as a novel marker of all-cause mortality. J Am Soc Nephrol. 2015 Jun;26(6):1426-33. doi: 10.1681/ASN.2014010115. Epub 2014 Oct 24. PMID 25343954
- [Background] Schmieder RE, Messerli FH, Garavaglia G, Nunez B. Glomerular hyperfiltration indicates early target organ damage in essential hypertension. JAMA. 1990 Dec 5;264(21):2775-80. PMID 2146412
- [Background] Maeda I, Hayashi T, Sato KK, Koh H, Harita N, Nakamura Y, Endo G, Kambe H, Fukuda K. Cigarette smoking and the association with glomerular hyperfiltration and proteinuria in healthy middle-aged men. Clin J Am Soc Nephrol. 2011 Oct;6(10):2462-9. doi: 10.2215/CJN.00700111. Epub 2011 Sep 1. PMID 21885794
- [Background] Melsom T, Mathisen UD, Eilertsen BA, Ingebretsen OC, Jenssen T, Njolstad I, Solbu MD, Toft I, Eriksen BO. Physical exercise, fasting glucose, and renal hyperfiltration in the general population: the Renal Iohexol Clearance Survey in Tromso 6 (RENIS-T6). Clin J Am Soc Nephrol. 2012 Nov;7(11):1801-10. doi: 10.2215/CJN.02980312. Epub 2012 Aug 23. PMID 22917703
- [Background] Mogensen CE, Christensen CK. Predicting diabetic nephropathy in insulin-dependent patients. N Engl J Med. 1984 Jul 12;311(2):89-93. doi: 10.1056/NEJM198407123110204. PMID 6738599
- [Background] Benz K, Amann K. Maternal nutrition, low nephron number and arterial hypertension in later life. Biochim Biophys Acta. 2010 Dec;1802(12):1309-17. doi: 10.1016/j.bbadis.2010.03.002. Epub 2010 Mar 10. PMID 20226855
- [Background] Sethi S, D'Agati VD, Nast CC, Fogo AB, De Vriese AS, Markowitz GS, Glassock RJ, Fervenza FC, Seshan SV, Rule A, Racusen LC, Radhakrishnan J, Winearls CG, Appel GB, Bajema IM, Chang A, Colvin RB, Cook HT, Hariharan S, Herrera Hernandez LP, Kambham N, Mengel M, Nath KA, Rennke HG, Ronco P, Rovin BH, Haas M. A proposal for standardized grading of chronic changes in native kidney biopsy specimens. Kidney Int. 2017 Apr;91(4):787-789. doi: 10.1016/j.kint.2017.01.002. PMID 28314581
- See also: Homepage Clinical Research Center — https://www.medizin4.uk-erlangen.de/forschung/klinische-forschungsstation-crc/